CLINICAL TRIAL: NCT01543659
Title: A Phase I/II Study of Clinical and Molecular Correlates of Positron Emission Tomography (PET) With 89Zr-DFO-huJ591 in Metastatic Prostate Cancer
Brief Title: Clinical and Molecular Correlates of Positron Emission Tomography (PET) With 89Zr-DFO-huJ591 in Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); Broad Institute of MIT and Harvard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-126
Record Dates: First submitted 2012-02-22; First posted 2012-03-05 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: 89Zr-DFO-huJ591; prostate; Pet scan; 11-126
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Laboratories

ARMS (1):
- 89Zr-DFO-huJ591 (Experimental): Registered patients will undergo a baseline FDG PET scan up to 14 days before administration of a single dose of the 89Zr-DFO-huJ591 tracer, this scan is considered for research purposes. The exception to the 14-day timeframe is that patients who have already had an FDG PET scan up to 4 weeks prior to registration are not required to repeat the FDG PET scan on study.
  Interventions: Drug: 89Zr-DFO-huJ591

INTERVENTIONS:
Drug: 89Zr-DFO-huJ591 — The first 10 patients enrolled in the study will undergo serial whole-body scans to allow assessment of 89Zr-DFO-huJ591 biodistribution. There will be no intervening changes in therapy between the scans. The first 10 patients enrolled will also have serial blood samples drawn for PK analysis (2 -3 mL per time point). The remaining 90 patients enrolled (Patients 11-100) will have only 1 whole-body scan, at a time point to be determined based on the results for the first 10 patients. Biopsies are not mandatory, but highly recommended for the scientific purposes of the study. If feasible and the patient consents, all patients will undergo either or both of the following: (a) core biopsy of soft tissue site of disease; (b) core biopsy of bony site of disease. These biopsies will be performed following the last whole-body scan, prior to initiation of a new intervening therapy, and no more than 4 weeks after 89Zr-DFO-huJ591 administration.
  Other Names: Tissue will be analyzed for AR axis genomic and proteomic pathways by Dr. Loda's; laboratory.

SUMMARY:
The purpose of this study is to define the safety and accuracy of 89Zr-DFO-huJ591 PET scans. By improving our ability to find cancer cells, the investigators hope to be able to improve treatment for patients in the future.

The study doctors want to determine whether a new kind of scan, called a 89Zr-DFO-huJ591 PET scan, can specifically see prostate cancer that has spread to other parts of the body, especially the bones. The study doctors will also look at how the 89Zr-DFO-huJ591 reacts with the body and how long it stays in the body. The investigators will also ask the patient to have a biopsy performed. The study doctors will compare the findings the investigators see on the scans with findings on the optional tissue biopsy. Finally, the investigators will compare the pictures from a 89Zr-DFO-huJ591 PET scan with those of a standard PET scan (called FDG PET) and standard CT scans or magnetic resonance (MRI) scans or bone scans, depending on which standard scans the doctor has ordered.

PET scanning uses a small amount of radiation attached to a molecule that is taken up by the cancer. In this trial, the patient will undergo two types of PET scans. One uses FDG. FDG is a standard tracer for PET scans. The patient will also undergo another type of PET scan that is experimental. This experimental PET uses a radioactive protein called J591. The radiation source is a type of metal called zirconium-89 (89Zr). The whole tracer, J591 plus the 89Zr, is abbreviated as 89Zr-DFO-huJ591. This tracer is what is being studied. The tracer used in a scan should find where the cancer is in the body.

ELIGIBILITY:
Inclusion Criteria:

Metastatic Prostate Cancer Patients:

* Adult male ≥ 18 years of age
* Patients with histologically confirmed prostate cancer at MSKCC
* Progressive disease manifest by either:
* Imaging modalities:
* Bone Scan: New osseous lesions on bone scan and/or
* MRI or CT: An increase in measurable soft tissue disease or the appearance of new sites of disease.

OR

* Biochemical progression:

At least 3 rising PSA values from a baseline that are obtained 1 week or more apart, or 2 measurements obtained 2 or more weeks apart. The increase over the range of values should be at least 25%.

* Visible lesions by CT, bone scan, or MRI that are consistent with disease
* Performance status of 60 or higher (Karnofsky scale) (Appendix B)
* Ability to understand and willingness to sign a written informed consent document

Rising PSA Prostate Cancer Patients:

* Adult male ≥18 years of age
* Patients with histologically confirmed prostate cancer at MSKCC
* Undergone radical prostatectomy
* Detectable PSA (>0.05 ng/mL) that rises on subsequent evaluation
* Radiographic evaluation involving bone imaging and cross sectional imaging of at least the pelvis that is negative or equivocal for metastatic disease
* Performance status of 60 or higher (Karnofsky scale) (Appendix B)
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients meeting any of the following criteria will not be eligible for study entry (Metastatic and Rising PSA cohorts):
* Previous anaphylactic reaction to either J591 or FDG
* Hepatic laboratory values
* Bilirubin > 1.5 x ULN (institutional upper limits of normal) Exception: patient's with a history of Gilbert's disease
* AST/ALT > 2.5 x ULN
* Albumin < 2 g/dL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
ability of 89Zr-DFO-huJ591 PET to detect known sites of disease | 3 years
  With 50 patients enrolled over 3 years and an anticipated 20 lesions per patient, our estimate of sensitivity will be based on approximately 1000 lesions. Assuming an intra-patient correlation of 0.1 (based on our experience of FDG PET in this disease) we will be able to estimate the sensitivity within ±9% of its true value, assuming that the true sensitivity is 50%. If the sensitivity is higher then our estimates will be more precise. The findings from the optimal scan of 89Zr-DFO-huJ591 PET in the first 10 patients will be used for this purpose.
the pharmacokinetics (PK) and biodistribution of 89Zr-DFO-huJ591 PET | 3 years
  For the first 10 patients, 89Zr-DFO-huJ591 PET scan will be repeated on Days 2, 3-6, and 7-8 based on a single injection given at Day 1. The uptake from these subsequent scans will be used to determine the pharmacokinetics and the biodistribution of 89Zr-DFO-huJ591 as a function of time from injection. Pharmacokinetic analysis will be performed using a biexponential model non-compartmental analysis; standard parameters such as AUC, clearance, volume of distribution, Tmax, and Cmax will be reported.

SECONDARY OUTCOMES:
To use 89Zr-DFO-huJ591 PET image guided biopsies as a means for improved sampling of individual lesions of metastatic prostate cancer | 3 years
  The hit rate, defined as presence of tumor in the biopsied lesion, will be compared with the historical control of 25% (which is the estimated hit rate of FDG PET from our previous studies). Based on historical experience in this patient population we anticipate that we will obtain 33 biopsied lesions (an average contribution of 1 biopsied lesion from 33 consenting patients), which will provide approximately 80% power to distinguish hit rates of 25% and 45% (one-sample two-sided binomial test controlling Type I error at 5%).
PSMA and AR expression and AR axis genomic and proteomic pathways on tumor tissue with the 89Zr-DFO-huJ591 PET imaging characteristics | 3 years
  89Zr-DFO-huJ591 uptake will be compared by PSMA and AR expression on tumor tissues (present/absent) using the rank-sum test. Results will also be presented using side-by-side histograms and box plots.
FDG PET with 89Zr-DFO-huJ591 PET tumor uptake | 3 years
  All lesions with uptake will be used to correlate the accumulation of 89Zr-DFO-huJ591 to FDG. The width of the estimated confidence interval as a function of the value of the correlation coefficient (ρ) are given in Table 3. This assumes that uptake is normally distributed and for planning purposes only. Actual data analysis will make use of the rank correlation. These values conservatively assume a single lesion per patient. With multiple lesions per patient, narrower confidence intervals will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/